CLINICAL TRIAL: NCT05097092
Title: Strength Training Augmenting Rehabilitation - 1
Brief Title: Strength Training Augmenting Rehabilitation
Acronym: STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Joshua Carr, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-101
Record Dates: First submitted 2021-09-22; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Muscle Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilization control (Experimental): The immobilization control group will undergo arm immobilization. Immobilization will be implemented with four weeks of muscle unloading with a sling and swathe on the nondominant arm. The sling will suspend the arm at the elbow joint with the elbow in a flexed position at 90°, the swathe will then wrap around the participant to fix the arm against the body.
  Interventions: Procedure: Orthopedic immobilization; Other: Bilateral resistance training
- Immobilization with unilateral training (Experimental): The immobilization with unilateral training group will undergo arm immobilization for four with a sling and swathe on the nondominant arm. The sling will suspend the arm at the elbow joint with the elbow in a flexed position at 90°, the swathe will then wrap around the participant to fix the arm against the body. The free (non-immobilzed) arm of this group will undergo heavy strength training twice per week throughout the immobilization period. The training will consist of unilateral dumbbell shoulder press and biceps curl.
  Interventions: Procedure: Orthopedic immobilization; Other: Unilateral resistance training; Other: Bilateral resistance training

INTERVENTIONS:
Procedure: Orthopedic immobilization — Orthopedic immobilization will be performed with a sling and swathe.
Other: Unilateral resistance training — Unilateral resistance training will be performed by the dominant arm of the immobilization + unilateral resistance training group during Phase 1.
  Arms: Immobilization with unilateral training
Other: Bilateral resistance training — Bilateral resistance training will be performed by both arms in both groups during Phase 2.

SUMMARY:
This project aims to determine whether a novel strength training rehabilitation protocol can diminish the negative consequences of limb immobilization and expedite the restoration of muscle function during retraining in healthy individuals.

DETAILED DESCRIPTION:
The present study will examine the time course of muscle strength and size adaptations in two groups of volunteers during immobilization and retraining. Both groups will undergo temporary muscle disuse by wearing a shoulder sling and swathe on their non-dominant arm for ~≥10 hours/day for four weeks. One group (immobilization + unilateral training) will perform progressive unilateral strength training of the free limb throughout the immobilization period. The other group (immobilization control) will not undergo any training during the immobilization period. Following immobilization, both groups will undergo four weeks of bilateral strength training to retrain the immobilized arm.

ELIGIBILITY:
Inclusion Criteria:

* a body mass index between 18 - 35 kg/m2
* 18-35 years of age
* right-hand dominant
* willingness to comply with the immobilization requirements
* willingness to refrain from strength training outside of the study
* willingness to comply with the strength training procedures of the study

Exclusion Criteria:

* a personal or family history of blood clots
* a personal or family history of thyroid disorders
* previous orthopedic surgeries to the upper limbs and/or joint pain of the upper limbs in the last 6 months
* neuromuscular or metabolic disorders
* osteoarthritis
* use of hormone replacement therapy (ie., testosterone, estrogen, and/or growth hormone pharmaceuticals)
* pregnancy and/or nursing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-08-13 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
Changes in isometric muscle strength | Changes from baseline at 5 and 10 weeks
  MVC (Newton)
Changes in dynamic muscle strength | Changes from baseline at 5 and 10 weeks
  1RM (lbs)
Changes in muscle size | Changes from baseline at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 weeks
  Ultrasound muscle thickness of biceps brachii and triceps brachii
Changes in lean mass | Changes from baseline at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 weeks
  DEXA
Changes in EMG amplitude | Changes from baseline at 5 and 10 weeks
  Surface EMG
Changes in action potential amplitude | Changes from baseline at 5 and 10 weeks
  Surface EMG Decomposition

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TCU Neuromuscular Physiology Laboratory, Fort Worth, Texas
  - TCU RIC, Fort Worth, Texas